CLINICAL TRIAL: NCT07404527
Title: Usefulness of Bioelectrical Impedance Analysis for Perioperative Fluid Evaluation and Complication Prediction in Oncological Patients Undergoing Colorectal Surgery
Brief Title: Bioelectrical Impedance Analysis for Perioperative Fluid Evaluation in Colorectal Cancer Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Oncology Ljubljana (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: OI-2023-BIA; ERIDNPVO-0070/2023 (Other: Ethics Committee of the Institute of Oncology Ljubljana)
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Gastrointestinal Cancer; Digestive System Neoplasms
Keywords: SARC-F
MeSH Terms: conditions — Gastrointestinal Neoplasms; Digestive System Neoplasms | interventions — Cetuximab

STUDY DESIGN:
Intervention Model Description: Single-group study assessing sarcopenia risk using the SARC-F screening tool at baseline and during systemic treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): Patients receive induction chemotherapy followed by chemoradiotherapy with cetuximab.
  Interventions: Drug: Cetuximab (CRC)

INTERVENTIONS:
Drug: Cetuximab (CRC) — Cetuximab is administered in combination with induction chemotherapy followed by concurrent chemoradiotherapy, according to the study protocol.

SUMMARY:
Sarcopenia is a complex syndrome characterized by progressive and generalized loss of skeletal muscle mass and strength. In patients with cancer, sarcopenia is associated with poorer prognosis, increased treatment-related toxicity, higher postoperative complication rates, reduced response to therapy, and decreased quality of life. Importantly, sarcopenia may be present even in patients with preserved nutritional status or overweight.

Patients with gastrointestinal cancers are at particularly high risk of developing sarcopenia, both as a consequence of the malignant disease itself and as a result of systemic anticancer treatment. Early identification of patients at risk is therefore essential in order to enable timely nutritional and supportive interventions.

The aim of this study is to evaluate the proportion of patients with gastrointestinal cancer who screen positive for sarcopenia risk using the SARC-F questionnaire before the start of systemic treatment and during treatment. Patients with a positive screening result will be referred for further clinical nutritional assessment and managed according to a multidisciplinary approach.

DETAILED DESCRIPTION:
Sarcopenia is recognized as an important negative prognostic factor in oncology, independent of malnutrition. It contributes to increased morbidity and mortality, higher incidence of treatment-related toxicity, reduced tolerance to systemic therapy, and impaired functional status. In patients with gastrointestinal malignancies, sarcopenia is common due to tumor-related metabolic changes, reduced intake, inflammation, and the adverse effects of anticancer therapies.

The SARC-F questionnaire is a simple, validated screening tool recommended by the European Working Group on Sarcopenia in Older People (EWGSOP2) for the identification of individuals at risk of sarcopenia. It consists of short, function-oriented questions assessing strength, assistance in walking, rising from a chair, climbing stairs, and falls. A SARC-F score of ≥4 indicates increased risk of sarcopenia.

This prospective interventional study will include adult patients with gastrointestinal cancer who are candidates for systemic anticancer treatment. Participants will complete the SARC-F questionnaire at baseline, prior to initiation of systemic therapy, and again during treatment. The primary objective is to determine the proportion of patients with positive SARC-F screening results at these time points and to evaluate changes in sarcopenia risk during the course of treatment.

Patients who screen positive for sarcopenia risk will be referred to the clinical nutrition outpatient clinic for further assessment, including anthropometric measurements and, where clinically indicated, dual-energy X-ray absorptiometry (DXA). Based on the results, individualized multimodal interventions for the prevention and treatment of sarcopenia will be initiated in collaboration with a multidisciplinary team.

The study does not impose additional diagnostic or therapeutic burden beyond standard clinical care. The results are expected to contribute to improved early identification and management of sarcopenia in patients with gastrointestinal cancer.

ELIGIBILITY:
Inclusion Criteria:

Adult patients (≥18 years of age).

Histologically confirmed head and neck cancer.

Indication for induction chemotherapy followed by chemoradiotherapy with cetuximab.

Adequate organ function as required by the study protocol.

Ability to provide informed consent.

Exclusion Criteria:

* Prior systemic therapy or radiotherapy for head and neck cancer.

Presence of uncontrolled comorbidities that would preclude study treatment.

Known hypersensitivity to cetuximab or components of the treatment regimen.

Pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-10-24 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | Up to 5 years
  Overall survival is defined as the time from study enrollment to death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Oncology Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No